CLINICAL TRIAL: NCT05300958
Title: Deferoxamine Plus Chemotherapy for Metastatic Triple Negative Breast Cancer: A Single-armed, Phase II Trial
Brief Title: Deferoxamine Plus Chemotherapy for Metastatic Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty accruing subjects the study accrual was closed.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-017
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer
Keywords: Deferoxamine plus chemotherapy; Objective Response Rate and safety
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Deferoxamine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Deferoxamine：50mg/kg+500ml normal saline (NS) plus chemotherapy
  Interventions: Drug: Deferoxamine Plus Chemotherapy

INTERVENTIONS:
Drug: Deferoxamine Plus Chemotherapy — Deferoxamine：50mg/kg+500ml normal saline (NS)
  Other Names: Chemotherapy：Treatment of Physician's Choice (TPC)

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of chemotherapy plus deferoxamine in metastatic breast cancer whose evaluation is stable disease with a trend of progression.

DETAILED DESCRIPTION:
This is a phase II, single center, prospective, single arm clinical trial. A lot of in vitro and in vivo study demonstrate that deferoxamine can increase anti-tumor effect. The objective of the study is to evaluate the efficacy and safety of chemotherapy plus deferoxamine in metastatic breast cancer whose evaluation is stable disease with a trend of progression after second-line. This study plans to recruit 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Has measurable metastatic triple-negative breast cancer, with at least 1 measurable lesion per RECIST criteria.
* Fail second-line or above anti-tumor treatment
* Evaluation is stable disease with a trend of progression.
* Minimum life expectancy 16 weeks
* Histological confirmation of breast cancer on primary tumour at diagnosis/on biopsy of metastasis
* ECOG Performance Status (PS) 0-2 with no deterioration over previous 2 weeks
* Normal organ function.
* Has signed a Patient Informed Consent Form.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) score of ≥ 2
* Patients with severe liver and kidney insufficiency
* Deferoxamine Ingredients allergy
* With the exception of alopecia, any unresolved toxicities from previous therapy greater than CTCAE grade 1 before study treatment
* Inability or unwillingness to comply with study procedures, including inability to take regular oral medication
* Researchers consider it is not suitable for participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period

SECONDARY OUTCOMES:
clinical benefit rate (CBR) | 6 months
  the proportion of patients with tumors complete response, partial response, and stable disease
progression-free survival (PFS) | 6 months
  the time from the beginning of treatment for metastatic breast cancer to disease progression or death from any cause
overal survival (OS) | 12 months
  the time from the beginning of treatment for metastatic breast cancer to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-yu Yuan, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China